CLINICAL TRIAL: NCT00924196
Title: Natural History Study and Longitudinal Assessment of Children, Adolescents, and Adults With Neurofibromatosis Type 1
Brief Title: Natural History Study of Patients With Neurofibromatosis Type I
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080079; 08-C-0079; NCT00693394 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-08-21

CONDITIONS: Neurofibromatosis Type 1; Malignant Peripheral Nerve Sheath Tumor; Plexiform Neurofibroma; Optic Glioma; Neurofibroma
Keywords: Plexiform Neurofibroma; Optic Pathway Tumor; Neurofibroma; Malignant Peripheral Nerve Sheath Tumor; Volumetric MRI; Natural History; Neurofibromatosis Type 1; NF1; Optic Glioma
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibrosarcoma; Neurofibroma, Plexiform; Optic Nerve Glioma; Neurofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biologic parents of children and adults with NFI: Biologic parents of children and adults with NFI will be evaluated at one time point, using a Neuropsychological Test Battery and QOL Assessment. Closed to enrollment
- Children and adults with NFI: Children and adults with NFI whose tumor and non tumor related manifestations will be longitudinally evaluated. Closed to enrollment
- Unaffected siblings of children and adults with NFI: Unaffected siblings of children and adults with NFI will be evaluated at one time point using a Neuropsychological Test Battery and QOL Assessment. Closed to enrollment

SUMMARY:
Background:

Neurofibromatosis Type 1 (NF1) is a genetic disorder in which patients are at increased risk of developing tumors (usually non-cancerous) of the central and peripheral nervous system. The disease affects essentially every organ system.

The natural course of NFI over time is poorly understood. For most patients the only treatment option is surgery. A better understanding of NF1 may be helpful for the design of future treatment studies.

Objectives:

To evaluate people with NF1 over 10 years in order to better understand the natural history of the disease.

To characterize the patient population and to examine how NFI affects patients quality of life and function.

Eligibility:

Children, adolescents, and adults with NF1.

Design:

Participants have a comprehensive baseline evaluation including genetic testing, tumor imaging, pain and quality-of-life assessments, and neuropsychological, motor and endocrine evaluations.

Patients are monitored every 6 months to every 3 years, depending on their individual findings at the baseline study. Tests may include the following, as appropriate:

* Medical history, physical examination and blood tests.
* Whole body and face photography to monitor visible deformities.
* Neuropsychological testing, quality-of-life evaluations, motor function tests, endocrinologic evaluations, heart and lung function tests, hearing tests, bone density scans and other bone evaluations.
* MRI and PET scans to detect and assess plexiform neurofibromas (tumors that arise from nerves and can cause serious problems), paraspinal neurofibromas (tumors that arise from nerves around the spine and can cause problems by compressing the spinal cord), and malignant peripheral nerve sheath tumors (a type of cancer that arises from a peripheral nerve or involves the sheath covering the nerve).
* Eye exams, MRI scans and PET scans to evaluate optic pathway gliomas (tumors arising from the vision nerves or the brain areas for vision) and the chemicals within the tumor and brain.
* Eye exams and photographs to evaluate the development of Lisch nodules (non-cancerous tumors on the eye).
* Photographs of dermal neurofibromas (tumors of the skin), cafe-au-lait spots (dark or pigmented areas on the skin that are often the first signs of NF1) and other skin problems.
* Pain evaluations to monitor the different types of pain patients experience, causes of the pain, how often the pain occurs, effect of the pain on quality of life, and what pain medications and alternative treatments, such as acupuncture, are effective....

DETAILED DESCRIPTION:
Background

Neurofibromatosis Type 1 (NF1) is an autosomal dominant, progressive genetic disorder characterized by diverse clinical manifestations. Patients with NF1 have an increased risk of developing tumors of the central and peripheral nervous system including plexiform neurofibromas (PN), dermal neurofibromas, optic pathway tumors, brain tumors, malignant peripheral nerve sheath tumors (MPNST), juvenile myelomonocytic leukemia, and pheochromocytomas. In addition, NF1 manifests in essentially every organ system, with for example, skeletal and vascular abnormalities, and cognitive deficits. Thus, the care for individuals with NF1 requires a multidisciplinary approach. The natural history of NF1 related tumor and other manifestations is poorly understood, and for most NF1 related tumor manifestations the only standard treatment option is surgery. The NIH Clinical Center provides the ideal infrastructure for evaluation of the natural history of rare diseases. A better understanding of the natural history of NF1 related tumor and other manifestations will be helpful for the design of treatment studies. The NCI, POB has an active clinical trials program for NF1 related tumor manifestations including PN, MPNST. Unlike individuals with refractory solid cancers, individuals with NF1 have near normal life expectancy, and their benign tumors progress more slowly than solid cancers. Individuals with NF1 may thus participate in multiple treatment trials.

Objectives

The overall purpose of this descriptive NF1 Natural History study is to serve as an umbrella protocol for the ongoing NF1 clinical trials program to allow the longitudinal evaluation of individuals with NF1 for NF1 related tumor and non tumor manifestations irrespective whether they are currently enrolled on a treatment study or not, and to develop a better understanding of the biology of NF1 related manifestations. Following these patients longitudinally will allow investigators to develop a better understanding of the natural history of these manifestations, provide the basis for the development of endpoints for clinical trials and to potentially develop more effective treatments. NF1 manifestations, which will be followed longitudinally, include PN, MPNST, optic pathway tumors, dermal neurofibromas, NF1 associated pain, and neuropsychological, motor, and endocrine function. Patient samples will be collected to investigate the existence of a peripherally detectable disease progression biomarker. A comprehensive treatment plan and recommendations will be developed and communicated with the patient and primary caregivers.

Eligibility

Children, adolescents, and adults with a confirmed clinical diagnosis of NF1 or a confirmed NF1 mutation.

Design

Attempts will be made to have all individuals undergo a comprehensive baseline evaluation including clinical phenotyping, genotyping, imaging of tumor manifestations, and pain, quality of life, neuropsychological, motor, and endocrine evaluations. The NF1 manifestations will be longitudinally monitored with a frequency of every year to every three years, with the extent and timing of follow-up evaluations depending on the findings at baseline.

ELIGIBILITY:
* ELIGIBILITY CRITERIA PATIENT

INCLUSION CRITERIA:

1. Age:

   * Less than or equal to 35 years of age for new patients evaluated at NIH.
   * No upper age limit for patients previously enrolled on clinical trials at NIH or for patients diagnosed with MPNST, or with clinical concern for MPNST, or with infrequent or unusual NF1 related manifestations.
2. Diagnosis: Patients who are diagnosed with NF1 using the NIH Consensus Conference criteria or have a confirmed NF1 mutation with analysis performed in a CLIA-certified laboratory. NF1 mutation testing to confirm eligibility will not be performed on this protocol, but as part of a separate screening study. Histologic confirmation of NF1 related benign tumors is not necessary in the presence of consistent clinical and radiographic findings, but is required for individuals with MPNST who enroll on this study.

   For the clinical diagnosis of NF1 all study subjects must have at least two or more diagnostic criteria for NF1 listed below (NIH Consensus Conference):
   1. Six or more cafe-au-lait spots (greater than or equal to 0.5 cm in prepubertal subjects or greater than or equal to 1.5 cm in postpubertal subjects).
   2. Greater than or equal to 2 neurofibromas or 1 plexiform neurofibroma.
   3. Freckling in the axilla or groin.
   4. Optic glioma.
   5. Two or more Lisch nodules.
   6. A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex).
   7. A first-degree relative with NF1.
3. Prior and current therapy: For NF1 related benign tumor manifestations there is no standard effective medical treatment, and surgery is the only standard treatment. Chemotherapy and radiation therapy are additional treatment options for malignant NF1 related tumors. For the purpose of this study, subjects who have not previously received medical or surgical treatment, patients, who have previously received medical or surgical treatment, and patients who are currently receiving medical treatment and/or radiation for a NF1 related manifestation will be eligible. Prior and current treatment for NF1 related manifestations will be recorded at trial entry and throughout the study.
4. Performance Status: ECOG less than or equal to 3. Subjects who are wheelchair bound because of paralysis will be considered ambulatory when they are up in their wheelchair. Subjects have to be able to travel to the NIH for evaluations.
5. Informed Consent: All patients or their legal guardians (if the patient is less than 18 years old) must sign an IRB-approved document of informed consent to demonstrate their understanding of the investigational nature and the risks of this study before any protocol-related studies are performed. When appropriate, pediatric subjects will be included in all discussions.

EXCLUSION CRITERIA:

1. In the opinion of the investigator the patient is not able to return for follow-up visits or obtain required follow-up studies.
2. In the opinion of the investigator the patient is not able to obtain an MRI scan.
3. Individuals who are pregnant or breast feeding or who become pregnant while enrolled on this trial will not be excluded from participation, but will not undergo radiographic evaluations or MRI scans requested for research purposes, or other studies which might negatively impact on the pregnancy.

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a confirmed clinical diagnosis of NF1 or a confirmed NF1 mutation; unaffected siblings and biologic parents of the individuals with NFI who enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2008-02-25 (Actual)

PRIMARY OUTCOMES:
To serve as an umbrella protocol for the ongoing NF1 clinical trials program to longitudinally characterize and analyze NF1 related tumor and non-tumor manifestations, and to develop a better understanding of the biology of NF1 related manifesta... | throughout the study
  Characterized features will be described and presented.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Ferner RE. Neurofibromatosis 1 and neurofibromatosis 2: a twenty first century perspective. Lancet Neurol. 2007 Apr;6(4):340-51. doi: 10.1016/S1474-4422(07)70075-3. PMID 17362838
- [Background] Korf BR. Clinical features and pathobiology of neurofibromatosis 1. J Child Neurol. 2002 Aug;17(8):573-7; discussion 602-4, 646-51. doi: 10.1177/088307380201700806. PMID 12403555
- [Background] Kim A, Gillespie A, Dombi E, Goodwin A, Goodspeed W, Fox E, Balis FM, Widemann BC. Characteristics of children enrolled in treatment trials for NF1-related plexiform neurofibromas. Neurology. 2009 Oct 20;73(16):1273-9. doi: 10.1212/WNL.0b013e3181bd1326. PMID 19841379
- [Derived] Al Ghriwati N, Little P, Martin S, Tamula MA, Widemann BC, Wolters PL. Parent-child discrepancies in reports of child psychosocial functioning in neurofibromatosis type 1. J Fam Psychol. 2025 Feb;39(1):99-106. doi: 10.1037/fam0001256. Epub 2024 Oct 17. PMID 39418437
- [Derived] Curry BP, Alvarez R, Widemann BC, Johnson M, Agarwal PK, Lehky T, Valera V, Chittiboina P. Robotic Nerve Sheath Tumor Resection With Intraoperative Neuromonitoring: Case Series and Systematic Review. Oper Neurosurg. 2022 Feb 1;22(2):44-50. doi: 10.1227/ONS.0000000000000051. PMID 35007270
- [Derived] Akshintala S, Baldwin A, Liewehr DJ, Goodwin A, Blakeley JO, Gross AM, Steinberg SM, Dombi E, Widemann BC. Longitudinal evaluation of peripheral nerve sheath tumors in neurofibromatosis type 1: growth analysis of plexiform neurofibromas and distinct nodular lesions. Neuro Oncol. 2020 Sep 29;22(9):1368-1378. doi: 10.1093/neuonc/noaa053. PMID 32152628
- [Derived] Dagalakis U, Lodish M, Dombi E, Sinaii N, Sabo J, Baldwin A, Steinberg SM, Stratakis CA, Widemann BC. Puberty and plexiform neurofibroma tumor growth in patients with neurofibromatosis type I. J Pediatr. 2014 Mar;164(3):620-4. doi: 10.1016/j.jpeds.2013.10.081. Epub 2013 Dec 8. PMID 24321536
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0079.html